CLINICAL TRIAL: NCT03815357
Title: What is the Incidence of an Immune Disorder in Children With Invasive Pneumococcal Disease (IPD)? A Prospective Cohort Study.
Brief Title: What is the Incidence of an Immune Disorder in Children With Invasive Pneumococcal Disease (IPD)?
Status: Completed | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35266C
Record Dates: First submitted 2018-12-12; First posted 2019-01-24 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Invasive Pneumococcal Disease, Recurrent Isolated, 1; Invasive Pneumococcal Disease, Recurrent Isolated, 2; Invasive Pneumococcal Disease, Protection Against; Primary Immunodeficiency
Keywords: streptococcus pneumoniae; invasive pneumococcal disease; primary immunodeficiency
MeSH Terms: conditions — IRAK4 Deficiency; Invasive Pneumococcal Disease, Recurrent Isolated, 2; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with IPD: Children with IPD will be referred for immunological evaluation. The protocol for immune work up will be the same but between centres there is variation in the age criteria for referral i.e. >2 years in some, >6 months in others.
  Interventions: Other: Referral to Immunology

INTERVENTIONS:
Other: Referral to Immunology — Screening for primary immunodeficiency including splenic dysfunction

SUMMARY:
This is a multicentre prospective audit to determine the incidence of immunodeficiency in children with IPD.

Aims and/or research question of the project

1. To determine the incidence of primary immunodeficiency in children >2 years who present with IPD
2. To determine the types of immunodeficiency associated with IPD in children

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 18 years admitted to one of the six centres with IPD.

Exclusion Criteria:

* Children who do not fulfil the age criteria for immunological evaluation at that particular site e.g. aged <2 years at Royal Children's Hospital.
* Children with a known underlying condition predisposing to IPD i.e. nephrotic syndrome.

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children presenting with invasive pneumococcal disease at any of the participating sites listed.
  Invasive pneumococcal disease is defined by isolation by culture or PCR of Streptococcus pneumoniae from sterile sites including blood, cerebrospinal fluid (CSF), joint fluid or pleural fluid. In those patients with bacteraemia, their presentation needs to be accompanied by signs of sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
incidence of primary immunodeficiency in children who present with invasive pneumococcal disease | 3 years
  This will be picked up upon prospective immunological testing, after identification of patients with invasive pneumococcal disease. A series of tests will be performed depending on the clinical opinion of the immunology team. Such tests may include lymphocyte subsets, complement function, serum immunoglobulin levels, memory B cells, vaccine antibody responses, etc.
types of immunodeficiency associated with children who present with invasive pneumococcal disease | 3 years
  This will be determined based on the testing performed by the immunologists.

SECONDARY OUTCOMES:
whether increased referrals of children who present with invasive pneumococcal disease for investigation of primary immunodeficiency facilitates early detection | 3 years
  This information will come from reviewing the case series of patients who are identified from this study. The incidence of those with primary immunodeficiency will be analysed against known background rates of diagnoses.

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (5):
  - Sydney Children's Hospital, Sydney, New South Wales
  - Adelaide Women's and Children's Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Royal Children's Hospital, Melbourne, Victoria
  - Lady Cilento Children's Hospital, Brisbane
- Capital and Coast District Health Board, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaschignard J, Levy C, Chrabieh M, Boisson B, Bost-Bru C, Dauger S, Dubos F, Durand P, Gaudelus J, Gendrel D, Gras Le Guen C, Grimprel E, Guyon G, Jeudy C, Jeziorski E, Leclerc F, Leger PL, Lesage F, Lorrot M, Pellier I, Pinquier D, de Pontual L, Sachs P, Thomas C, Tissieres P, Valla FV, Desprez P, Fremeaux-Bacchi V, Varon E, Bossuyt X, Cohen R, Abel L, Casanova JL, Puel A, Picard C. Invasive pneumococcal disease in children can reveal a primary immunodeficiency. Clin Infect Dis. 2014 Jul 15;59(2):244-51. doi: 10.1093/cid/ciu274. Epub 2014 Apr 23. PMID 24759830
- [Background] Picard C, Puel A, Bustamante J, Ku CL, Casanova JL. Primary immunodeficiencies associated with pneumococcal disease. Curr Opin Allergy Clin Immunol. 2003 Dec;3(6):451-9. doi: 10.1097/00130832-200312000-00006. PMID 14612669
- [Background] Alsina L, Basteiro MG, de Paz HD, Inigo M, de Sevilla MF, Trivino M, Juan M, Munoz-Almagro C. Recurrent invasive pneumococcal disease in children: underlying clinical conditions, and immunological and microbiological characteristics. PLoS One. 2015 Mar 4;10(3):e0118848. doi: 10.1371/journal.pone.0118848. eCollection 2015. PMID 25738983